CLINICAL TRIAL: NCT05850936
Title: Effect of Medically Intraocular Pressure Lowering on Progressive High Myopia
Brief Title: Effect of IOP Lowering on Progressive HM
Acronym: PHM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiulan Zhang, Director of Clinical Research Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023KYPJ110
Record Dates: First submitted 2023-04-13; First posted 2023-05-09 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: High Myopia; Intraocular Pressure
Keywords: high myopia; intraocular pressure

STUDY DESIGN:
Intervention Model Description: Open-label, single-center, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Participants and physicians are not masked as to the treatment assignment. The study outcomes will be obtained by masked ophthalmic technicians according to standard protocols and read by masked graders at the End Point Adjudication Committee. The masking status of the technicians collecting data will be recorded at each study visit. The study data will be analyzed by masked researchers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): medical reduction of IOP by eyedrops
  Interventions: Drug: Assigned Interventions: IOP-lowering eye drops
- control arm (No Intervention): follow up without medication

INTERVENTIONS:
Drug: Assigned Interventions: IOP-lowering eye drops — IOP-lowering eye drops Xalacom eyedrops (combination drops, fixed latanoprost with timolol) will be the choice for treatment.
  Arms: Intervention arm

SUMMARY:
Currently, whether and when intraocular pressure (IOP) lowering medication should be used in progressive high myopia (HM) to control axial elongation is still a dilemma. Randomized trials are required to evaluate whether IOP lowering influences the growth of axial length in progressive HM eyes.

DETAILED DESCRIPTION:
Myopia has emerged as a major health issue in east Asia, especially the sight-threatening complications associated with high myopia (HM). Complication of HM can be associated with significant ocular morbidities including maculopathy, retinal detachment, and glaucoma.

Previous studies have shown that adult patients with HM have sustained growth of the axial length (AL), which is a risk factor for the progression of pathological myopia and thus may further affect the visual function , so how to slow down the sustained growth of the AL in adult patients with HM has become an urgent clinical problem. Previous studies have shown that IOP-lowering treatment is a protective factor for the growth of the AL in HM , and the results of animal experiments have further shown that medically IOP-lowering treatment can significantly slow down the AL lengthening and refractive changes in the guinea pig model of myopia. On this basis, the investigators proposed in a previous article that medically IOP-lowering treatment may slow down the growth of AL by three pathways related to the sclera and choroid: for the sclera, IOP-lowering treatment may reduce the scleral distending force, slow down the rate of scleral distension, and inhibit the activation of scleral fibroblasts to reduce scleral remodeling; for the choroid, IOP-lowering treatment may increase choroidal blood perfusion and for the choroid, hypotensive treatment can increase choroidal perfusion and thus reduce scleral remodeling due to scleral hypoxia. A previous retrospective study conducted by the investigators also shows that medically IOP-lowering treatment could control the progression of AL in HM, but there is still a lack of evidence from relevant robust randomized controlled clinical trials (RCT).

The investigators propose to conduct a RCT to evaluate whether medically IOP-lowering therapy is effective in controlling the progression of AL in HM. Secondly, this study also aims to provide data to evaluate IOP-lowering treatment effects on the incidence of changes in the visual field (VF), optic nerve head morphology including the retinal nerve fiber layer (RNFL), and retinal ganglion cell-inner plexiform layer (GC-IPL) loss, progression of myopic maculopathy, loss in visual function and change in quality of life. The outcomes of this study may provide a strong basis for treatment recommendations to control the progression of high myopic eyes, and to provide high-quality clinical research evidence for international clinical guidelines on myopia.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent given, and consent form signed.
2. Age between 18 and 65 years.
3. Diagnosed with HM: spherical equivalent ≤ -6.00 diopters or AL ≥ 26.5 mm.
4. Progressive HM: progression in AL ≥0.05mm in the past 6 months or ≥0.1mm in the past 12 months.
5. IOP ≥ 10 mmHg and ≤ 21mmHg on at least 2 visits, as measured by Goldmann applanation tonometry .
6. Best corrected visual acuity (BCVA) ≥ 6/12, and being able to obtain adequate AL examination, fundus photographs, optical coherence tomography (OCT) and complete the VF examination.

Exclusion Criteria:

1. Allergic to any kind of IOP-lowering therapy.
2. Combination of various serious fundus pathologies, such as proliferative diabetic retinopathy, retinal detachment, central retinal artery occlusion, etc.
3. Combination of chronic, recurrent or severe ocular inflammatory lesions, such as chronic or recurrent uveitis.
4. Patients with significant corneal or iris lesions, or severe cataract affecting fundus examination, or patients with only one eye.
5. Patients who have undergone any surgery or laser treatment affecting eye parameters during the follow-up period (within the last 1 year), such as cataract surgery.
6. Patients with other serious systemic diseases, such as hypertension, heart disease, diabetes, rheumatic immune system disease, etc., who cannot tolerate long-term follow-up and eye treatment.
7. Pregnant or lactating women, or those who plan to have children during the follow-up period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
progression of axial length (AL) | 12 months
  The number of subjects whose AL progressed during the follow up

SECONDARY OUTCOMES:
Incidence of visual field (VF) defects or progression | 12 months
  The number of subjects whose VF defects progressed during the follow up
Incidence of changes in the optic nerve head morphology including the retinal nerve fiber layer (RNFL) and ganglion cell-inner plexiform layer (GCIPL) | 12 months
  The number of subjects whose optic nerve head morphology including the RNFL and GCIPL changed during the follow up
progression of myopic maculopathy | 12 months
  The number of subjects whose myopic maculopathy progressed during the follow up

CONTACTS AND LOCATIONS:
Overall Officials: Xiulan Zhang, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leske MC, Hyman L, Hussein M, Heijl A, Bengtsson B. Comparison of glaucomatous progression between untreated patients with normal-tension glaucoma and patients with therapeutically reduced intraocular pressures. The effectiveness of intraocular pressure reduction in the treatment of normal-tension glaucoma. Am J Ophthalmol. 1999 May;127(5):625-6. No abstract available. PMID 10334369
- [Background] Garway-Heath DF, Crabb DP, Bunce C, Lascaratos G, Amalfitano F, Anand N, Azuara-Blanco A, Bourne RR, Broadway DC, Cunliffe IA, Diamond JP, Fraser SG, Ho TA, Martin KR, McNaught AI, Negi A, Patel K, Russell RA, Shah A, Spry PG, Suzuki K, White ET, Wormald RP, Xing W, Zeyen TG. Latanoprost for open-angle glaucoma (UKGTS): a randomised, multicentre, placebo-controlled trial. Lancet. 2015 Apr 4;385(9975):1295-304. doi: 10.1016/S0140-6736(14)62111-5. Epub 2014 Dec 19. PMID 25533656
- [Background] Leske MC, Heijl A, Hyman L, Bengtsson B. Early Manifest Glaucoma Trial: design and baseline data. Ophthalmology. 1999 Nov;106(11):2144-53. doi: 10.1016/s0161-6420(99)90497-9. PMID 10571351
- [Derived] Jiang J, Lin T, Lin F, Kong K, Wang P, Song Y, Zhou F, Wang Z, Jin L, Liu Y, Gao X, Chen J, Chen M, Lam DSC, Jonas JB, Chen S, Zhang X; Glaucoma Suspects with High Myopia Study Group. Effect of intraocular pressure reduction on progressive high myopia (PHM study): study protocol of a randomised controlled trial. BMJ Open. 2024 Jun 5;14(6):e084068. doi: 10.1136/bmjopen-2024-084068. PMID 38839388
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC11163624/